CLINICAL TRIAL: NCT04029766
Title: A Phase 1 Study to Investigate a Single Bolus Dose Followed With a 30 Minute Constant Infusion of HSK3486 on the Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of HSK3486 in Healthy Male Subjects.
Brief Title: A Study Evaluating Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of HSK3486 Single Bolus Dose Followed With a 30 Minute Constant Infusion in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK3486Australia-03
Record Dates: First submitted 2019-07-04; First posted 2019-07-23 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2019-06

CONDITIONS: Anesthesia; Sedation
MeSH Terms: interventions — HSK3486

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSK3486 (Experimental): 0.288 mg/kg bolus (1 min)+ 1 mg/kg/h constant infusion (30 min) or 0.540 mg/kg bolus (1 min)+ 2 mg/kg/h constant infusion (30 min)
  Interventions: Drug: HSK3486

INTERVENTIONS:
Drug: HSK3486

SUMMARY:
This study was a single center, open-label, single dose escalation study in healthy male subjects to investigate a bolus dose followed by a 30 minute constant infusion of HSK3486 over two cohorts.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male, aged 18 - 49 years (inclusive);
* 2. Be in general good health without clinically significant medical history;
* 3. American Society of Anesthesiologists (ASA) Physical Status Classification of I or II;
* 4. Body Mass Index (BMI) between 18 and 30 kg/m2 (inclusive);
* 5. Negative screen for drugs of abuse, alcohol, hepatitis B surface antigen (HBs-Ag), hepatitis C (HCVAb) and Human Immunodeficiency Virus (HIV) at Screening; and drugs of abuse, alcohol pre dose on Day -1
* 6. Normal or non-clinically significant findings on a physical examination, 12-lead electrocardiogram (ECG) and vital signs (respiration rate between 12 and 20 breaths per minute, blood pressure (BP) between 100-140/60-90 mmHg, heart rate between 50-99 beats per minute, temperature between 35.8°C and 37.5°C and pulse oximetry values > 95% on room air.);
* 7. Clinical laboratory values within the normal limits as defined by the clinical laboratory, unless the Investigator decided that out-of-range values were not clinically significant;
* 8. Ability to provide written informed consent;
* 9. Willing and able to follow study instructions and likely to complete all study requirements;
* 10. Suitable venous and arterial access.

Exclusion Criteria:

* 1. History of allergy or sensitivity to: propofol, components of Fresofol 1% MCT/LCT propofol, or HSK3486 (excipients soy bean oil, glycerine, triglycerides, purified egg phospholipids, sodium oleate and sodium hydroxide), or plain lignocaine;
* 2. History of clinically significant problems with general anesthesia;
* 3. Current smoker, or a history of regular (more than weekly) use of tobacco- or nicotine-containing products within 2 months prior to Screening;
* 4. History of excessive alcohol intake (more than four standard drinks daily, on average) or use of recreational drugs within the last 3 months;
* 5. Use of prescription or over the counter medications within 7 days of Investigational Product administration, with the exception of contraceptive medications, paracetamol, oral non-steroidal antiinflammatory agents, topical over the counter preparations and routine vitamins (if they do not exceed an intake of 20 to 600 times the recommended daily dose), unless agreed as non-clinically relevant by the Principal Investigator and Sponsor;
* 6. Standard donation of blood within 30 days of the study;
* 7. Donation of plasma or participation in a plasmapheresis program within 7 days preceding this study;
* 8. Receipt of any investigational study drug within 30 days prior to Screening;
* 9. Unable to fast for the 6 hours prior to Investigational Product administration;
* 10. Clinically significant (as judged by the Investigator) presence of acute illness (e.g. gastrointestinal illness, infection such as influenza, upper respiratory tract infection) at admission to the clinical study unit;
* 11. Anticipated need for surgery or hospitalization during the study;
* 12. Anatomical abnormality that would potentially interfere with airway management under unconscious sedation or anesthesia;
* 13. History of posture-related gastric reflux more than twice weekly;
* 14. History of seizures or epilepsy ;
* 15. History of ischaemic heart disease;
* 16. History of brady- or tachy-dysrhythmias requiring medical care;
* 17. History of asthma, with bronchospasm requiring treatment in the last 3 months;
* 18. Any condition, which in the Investigator's opinion, put the subject at significant risk, could confound the study results or may interfere significantly with the subject's participation in the study.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2015-12-14 (Actual); Study Completion 2016-06-09 (Actual)

PRIMARY OUTCOMES:
Safety by measurement of Adverse Events | First dose of study drug on day 1

SECONDARY OUTCOMES:
Modified observer's assessment of alertness/sedation（MOAA/S） | From first dose of study drug until fully alert on day 1
  Observe the change of modified observer's assessment of alert /sedation during the whole trial
Bispectral index （BIS） | From first dose of study drug until fully alert on day 1
Median effective dose (ED50) | From first dose of study drug until fully alert on day 1
Peak concentration (Cmax) | From the start of administration to 48 hours after administration
Time to plasma peak concentration(Tmax) | From the start of administration to 48 hours after administration
Terminal elimination half life (t1/2z) and mean residence time (MRT) | From the start of administration to 48 hours after administration
Mean residence time (MRT) | From the start of administration to 48 hours after administration
Area Under the Curve (AUC0-30min, AUC0-1h, AUC0-last, and AUC0-inf) | From the start of administration to 48 hours after administration
Total clearance (CL) | From the start of administration to 48 hours after administration